CLINICAL TRIAL: NCT00916929
Title: Detect Fluid Early From Intra-thoracic Impedance Monitoring
Acronym: DEFEAT-PE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 40006062/D
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Implantable Cardioverter Defibrillator (ICD) (Other): Impedance Monitoring Feature in an Implantable Cardioverter Defibrillator (ICD).
  Interventions: Device: Impedance Monitoring Feature
- Cardiac Resynchronization Therapy (CRT-D) (Other): Impedance Monitoring Feature in a Cardiac Resynchronization Therapy (CRT-D) device.
  Interventions: Device: Impedance Monitoring Feature

INTERVENTIONS:
Device: Impedance Monitoring Feature — Algorithm in cardiac device that measures intra-thoracic impedance from the implanted leads

SUMMARY:
To demonstrate the safety and effectiveness of the Impedance Monitoring Feature in St Jude Medical cardiac devices.

ELIGIBILITY:
Inclusion Criteria:

* Must have a St. Jude Medical (SJM) ICD or CRT-D for at least 31 days
* Must have had an episode of acute decompensated heart failure (ADHF) within the past 6 months

Exclusion Criteria:

* History of kidney disease requiring hemodialysis
* Refractory end stage heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin K Heist, MD, PhD, Study Chair — Massachusetts General Hospital
Locations (34):
- United States (34):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Arkansas Cardiology, PA, Little Rock, Arkansas
  - Little Rock Cardiology Clinic, PA, Little Rock, Arkansas
  - Glendale Memorial Hospital and MC, Glendale, California
  - Cardiac Rhythm Specialists, Inc, Northridge, California
  - Colorado Cardiac Alliance, LLC, Colorado Springs, Colorado
  - Shands Jacksonville, Jacksonville, Florida
  - Watson Clinic Center, Lakeland, Florida
  - Orlando Heart Center, Orlando, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Iowa Heart Center, West Des Moines, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cardiology Consultants of East Michigan, Flint, Michigan
  - Thoracic Cardiovascular HC Found. (Sparrow Research), Lansing, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Associated Cardiovascular Consultants, Cherry Hill, New Jersey
  - New York Presbyterian Hospital / Cornell University, New York, New York
  - Mid Carolina Cardiology, Charlotte, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Mercy Hospital Fairfield, Fairfield, Ohio
  - Saint Vincent Consultants in Cardiovascular Diseases, Erie, Pennsylvania
  - Hospital of the University of PA, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - St Thomas Hospital, Nashville, Tennessee
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - The Hope Heart Institute, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient enrollment began on June 9, 2009 and ended on June 30, 2010. All patients had to be implanted at least 31 days prior to enrollment with a legally marketed St Jude Medical device capable of enabling the impedance monitoring feature.
Groups:
- Implantable Cardioverter Defibrillator (ICD) Device: Impedance Monitoring Feature: Implantable Cardioverter Defibrillator (ICD) algorithm measures impedance from 2 vectors: right ventricle to can and right ventricle to coil
- Cardiac Resynchronization Therapy (CRT-D) Device: Impedance Monitoring Feature: Cardiac Resynchronization Therapy device algorithm measures impedance from 2 vectors: left ventricle to can and right ventricle to coil.
Period: Overall Study
Arm/Group | Implantable Cardioverter Defibrillator (ICD) Device | Cardiac Resynchronization Therapy (CRT-D) Device
Started | 80 | 82
Completed | 70 | 53
Not Completed | 10 | 29
Not completed — Lost to Follow-up | 1 | 3
Not completed — Death | 5 | 10
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Left ventricular epicardial lead | 1 | 2
Not completed — Transferred to hospice care | 1 | 1
Not completed — System explant | 1 | 0
Not completed — Moved to another state | 0 | 1
Not completed — Device unable to process impedance data | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- ICD Device: Impedance Monitoring Feature: Implantable Cardioverter Defibrillator (ICD) algorithm measures impedance from 2 vectors: right ventricle to can and right ventricle to coil
- CRT-D Device: Impedance Monitoring Feature: Cardiac Resynchronization Therapy (CRT-D) algorithm measures impedance from 2 vectors: left ventricle to can and right ventricle to coil.
- Total: Total of all reporting groups
Arm/Group | ICD Device | CRT-D Device | Total
Number analyzed (Participants) | 80 | 82 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 36 | 80
  >=65 years | 36 | 46 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (14) | 66 (13) | 64 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 13 | 45
  Male | 48 | 69 | 117
Region of Enrollment [Number; unit: participants]
  United States | 80 | 82 | 162

OUTCOME MEASURES:

1. Primary Outcome: False Positive Rate
Description: False Positive Rate is the the number of departures from the device's programmed threshold that are unrelated to a heart failure event. The False Positive Rate per patient year of follow up should be less than 1.5.
Time Frame: 6-months
Population: All patients participating in the study were included in the analysis with a total of 82 patients in each arm. Of the 82 patients implanted with ICD, 2 were upgraded to CRT-D. These 2 patients were censored from the ICD cohort and included in the CRT-D cohort at the time of upgrade based on as-treated analysis principle resulting.
Measure: Number (95% Confidence Interval); unit: departures from device threshold
Groups:
- Cardiac Resynchronization Therapy (CRT-D) Device: Algorithm in cardiac device that measures intra-thoracic impedance from the implanted leads
- Implantable Cardioverter Defibrillator (ICD) Device: Algorithm in cardiac device that measures intra-thoracic impedance from implanted leads
Arm/Group | Cardiac Resynchronization Therapy (CRT-D) Device | Implantable Cardioverter Defibrillator (ICD) Device
Number analyzed (Participants) | 84 | 80
departures from device threshold | 1.8 [1.8 to 2.17] | 1.49 [1.49 to 1.8]
Statistical Analysis 1: Comparison: Cardiac Resynchronization Therapy (CRT-D) Device vs Implantable Cardioverter Defibrillator (ICD) Device; For each patient cohort, the hypothesis is formally expressed as follows: H0: Expected False Positive Rate ≥1.5 per patient-year of follow-up Ha: Expected False Positive Rate <1.5 per patient-year of follow-up The null hypothesis is rejected at the 5% significance level if the 95% upper confidence limit (UCL) for expected FPR is less than 1.5 per patient-year of follow-up; Test type: Superiority or Other; exact method; 95% Upper Confidence Limit of objective performance criteria; rate per patient year of follow up = 1.5

2. Secondary Outcome: Sensitivity
Description: Sensitivity is defined as the ability of the algorithm to detect heart failure events. Sensitivity is calculated as the number of heart failure events detected by the algorithm (true positives) divided by the total number of heart failure events (true positives + false positives).
Time Frame: 6-months
Population: All patients enrolled in the study were included in this analysis with a total of 82 patients in each group. Of the 82 patients implanted with ICD, 2 were upgraded to CRT-D during data collection period. These 2 patients were censored from ICD cohort and included in CRT-D cohort at the time of upgrade based on as-treated analysis principle.
Measure: Number (95% Confidence Interval); unit: percentage of true positives
Groups:
- Cardiac Resynchronizaiton Therapy (CRT-D) Device; Implantable Cardioverter Defibrillator (ICD) Device: Algorithm in cardiac device that measures intra-thoracic impedance from the implanted leads
Arm/Group | Cardiac Resynchronizaiton Therapy (CRT-D) Device | Implantable Cardioverter Defibrillator (ICD) Device
Number analyzed (Participants) | 84 | 80
percentage of true positives | 40 [26 to 40] | 30.8 [16.3 to 30.8]
Statistical Analysis 1: Comparison: Cardiac Resynchronizaiton Therapy (CRT-D) Device vs Implantable Cardioverter Defibrillator (ICD) Device; For each patient cohort, the hypothesis is formally expressed as follows: H0: Sensitivity ≤ 50% Ha: Sensitivity > 50% The desired outcome was to reject the null hypothesis at the 5% significance level. The null hypothesis is rejected at the 5% significance level if the 95% lower confidence limit (LCL) for sensitivity is greater than 50%; Test type: Superiority or Other; exact method; sensitivity = 50, 95% CI 1-sided [lower limit 50], Standard Error of Mean 5

ADVERSE EVENTS:
Time Frame: 755.98 patient months for CRT-D cohort; 902.37 patient months for ICD cohort
Arm/Group | CRT-D Device | ICD Device
Serious Adverse Events (participants affected / at risk) | 2/82 | 3/80
Other Adverse Events (participants affected / at risk) | 6/82 | 8/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT-D Device (N=82) | ICD Device (N=80)
Device Migration (Cardiac disorders) | 1 (1) | 0 (0)
Loss of Capture (LV lead related) (Cardiac disorders) | 1 (1) | 0 (0)
Lead dislodgement / migration (RV lead related) (Cardiac disorders) | 0 (0) | 1 (1)
Infection (system related) (Cardiac disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT-D Device (N=82) | ICD Device (N=80)
Elevated Pacing Threshold (LV lead related) (Cardiac disorders) | 1 (1) | 0 (0)
Phrenic Nerve / Diaphragmatic Stimulation (LV lead related) (Cardiac disorders) | 1 (1) | 0 (0)
Twiddler Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Therapy for Non Ventricular Rhythm (Cardiac disorders) | 3 (3) | 6 (8)
Bleeding / Hematoma (Cardiac disorders) | 0 (0) | 1 (1)
Unable to Turn Impedance Data Collection on (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There were no limitations of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less